CLINICAL TRIAL: NCT02029248
Title: National Study on the Quality of Life of Patients With Anorectal Malformation (MARQOL)
Brief Title: National Study on the Quality of Life of Patients With Anorectal Malformation
Acronym: MARQOL
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: MAREP ( Center For Rare Diseases Center Ano-Rectal And Pelvic Abnormalities) (Other)
Responsible Party: Sponsor
Other Study IDs: BRD/10/06-R
Record Dates: First submitted 2013-12-02; First posted 2014-01-07 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Anorectal Malformation
Keywords: Anorectal malformation; fecal incontinence; quality of life; child
MeSH Terms: conditions — Anorectal Malformations; Fecal Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Children 6-7: Patients who are between 6 and 7 years old
  Interventions: Other: Quality of life questionnaire
- Children 8-11: Patients who are between 8 and 11 years old
  Interventions: Other: Quality of life questionnaire
- Children 12-16: Patients who are between 12 and 16 years old
  Interventions: Other: Quality of life questionnaire
- Patients 17-30: Patients who are between 17 and 30 years old
  Interventions: Other: Quality of life questionnaire

INTERVENTIONS:
Other: Quality of life questionnaire

SUMMARY:
Anorectal malformations, occurring approximately 1 in 5000 live births, mainly involve the distal anus and rectum, but also sometimes the urinary and genital tracts. Defects range from the minor and easily treated with an excellent functional prognosis, to those that are complex and often associated with a poor functional prognosis.

Despite the better knowledge of the anatomy and physiology and the improvement of surgical management after birth, fecal and urinary incontinence can occur, due mainly to deficient nerve supply.

The quality of life of such patients is largely unknown in this country. The aim of the investigators study is to propose specific and generic questionnaires to the patients registered in the national database, correlated to their anatomical and functional status. A better understanding of such correlations should allow improvements in their medical and social management.

DETAILED DESCRIPTION:
Anorectal malformations (ARM), occurring approximately 1 in 5000 live births, mainly involve the distal anus and rectum, but also sometimes the urinary and genital tracts. Defects range from the minor and easily treated with an excellent functional prognosis, to those that are complex and often associated with a poor functional prognosis. Despite the better knowledge of the anatomy and physiology and the improvement of surgical management after birth, fecal and urinary incontinence can occur, due mainly to deficient nerve supply. A few studies and clinical practice have shown that disease-specific problems of ARM have an effect on somatic function, mental health and psychosocial functioning.

The assessment of quality of life requires a self-report questionnaire composed of items related to physical, emotional and social functioning, and disease-related symptoms. A specific ARM questionnaire, the HAQL, was developed by a Dutch team and published in 2001. Associated with generic questionnaire, it allowed quality of life assessment in Dutch population.

The quality of life of such patients is largely unknown in this larger country. The aim of the investigators study is to propose specific (HAQL translated from Dutch to French) and generic questionnaires to the patients registered in the national database, correlated to their anatomical and functional status.

A better understanding of such correlations should allow improvements in their medical and social management.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are between 6 and 30 years old
* Patients initially treated in a french pediatric surgery service for anorectal malformation

Exclusion Criteria:

* Patients lost from sight or dead
* Patients with concomitant malformations that can modify sphincter functions besides anorectal malformation (spina bifida, )
* Patients whose brain functions do not allow to reply to a questionnaire (mental retardation)

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients initially treated in a french pediatric surgery service for anorectal malformation
Sampling Method: Non-Probability Sample
Enrollment: 762 (Actual)
Dates: Start 2012-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Quality of life measured by HAQL specific questionnaire and two generic questionnaires: VSPA for children or WHOQOL-BREF for adults; functional status measured by Krickenbeck score | At the time of the inclusion
  HAQL: between 35 and 48 items (depending on the age of the patients) composing 8 dimensions; VSPA: 39 items composing 8 dimensions; WHOQOL-BREF: 26 items composing 4 dimensions; Krickenbeck: 3 items.

SECONDARY OUTCOMES:
Kind of malformation, associated malformation, sequelas, handicap degree, social integration | At the time of the inclusion
  Clinical questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Podevin, MD, PhD, Principal Investigator — CHU d'Angers (France)
Locations (37):
- France (37):
  - CHU Amiens, Amiens
  - CHU Angers, Angers
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - Hospices Civils de Lyon, Bron
  - CHU Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Hôpitaux Civils de Colmar, Colmar
  - CHU Dijon, Dijon
  - CHU Fort-de-France, Fort-de-France (Martinique)
  - CHU Grenoble, Grenoble
  - AP-HP Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - AP-HM La Timone, Marseille
  - AP-HM Hôpital Nord, Marseille
  - CHU Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHU Nice, Nice
  - CHR Orléans, Orléans
  - AP-HP Hôpital Trousseau, Paris
  - AP-HP Hôpital Necker, Paris
  - AP-HP Hôpital Robert Debré, Paris
  - CHU Pointe-à-Pitre, Pointe-à-Pitre (Guadeloupe)
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CHR La Réunion, Saint Denis (La Réunion)
  - CH Saint Brieuc, Saint-Brieuc
  - CHU Saint Etienne, Saint-Etienne
  - CHRU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHRU Tours, Tours
  - CHU Nancy, Vandœuvre-lès-Nancy

REFERENCES:
- [Background] Clermidi P, Podevin G, Cretolle C, Sarnacki S, Hardouin JB. The challenge of measuring quality of life in children with Hirschsprung's disease or anorectal malformation. J Pediatr Surg. 2013 Oct;48(10):2118-27. doi: 10.1016/j.jpedsurg.2013.03.071. PMID 24094967
- [Background] Mantoo S, Meurette G, Wyart V, Hardouin J, Cretolle C, Capito C, Sarnacki S, Podevin G, Lehur PA. The impact of anorectal malformations on anorectal function and social integration in adulthood: report from a national database. Colorectal Dis. 2013 Jun;15(6):e330-5. doi: 10.1111/codi.12186. PMID 23464709
- [Background] Podevin G, Petit T, Mure PY, Gelas T, Demarche M, Allal H, Becmeur F, Varlet F, Philippe P, Weil D, Heloury Y. Minimally invasive surgery for anorectal malformation in boys: a multicenter study. J Laparoendosc Adv Surg Tech A. 2009 Apr;19 Suppl 1:S233-5. doi: 10.1089/lap.2008.0137.supp. PMID 18973467
- [Background] Fleury J, Picherot G, Cretolle C, Podevin G, David A, Caillon J, Roze JC, Gras-le Guen C. Currarino syndrome as an etiology of a neonatal Escherichia coli meningitis. J Perinatol. 2007 Sep;27(9):589-91. doi: 10.1038/sj.jp.7211783. PMID 17724455